CLINICAL TRIAL: NCT06362720
Title: The Comparison the CMV Infection and Reactivation After Allogeneic Hematopoietic Stem Cell Transplantation Between Standard Regimen, Methotrexate Plus Cyclosporin A, and Post-transplant Cyclophosphamide-based Regimen
Acronym: CMV
Status: Not yet recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Chutima Kunacheewa, lecturer, Siriraj Hospital
Other Study IDs: 720/2566(IRB2)
Record Dates: First submitted 2024-04-03; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: CMV Infection or Reactivation After Allogenic HSCT
Keywords: CMV infection; CMV reactivation; allogenic HSCT; GVHD prophylaxis; posttransplant cyclophosphamide (PTCy); cyclosporin A; methotrexate
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard GVHD prophylaxis: calcineurin inhibitor (cyclosporin A ;CSA) and methotrexate (MTX)
- posttransplant cyclophosphamide (PTCy)

SUMMARY:
The goal of this observational study is to compare the CMV infection and reactivation after allogeneic hematopoietic stem cell transplantation Between Standard Regimen, Methotrexate plus Cyclosporin A, and Post-transplant Cyclophosphamide-based Regimen. The main questions it aims to answer are:

* How do CMV infection and reactivation differ between Allo-SCT patients who received a standard regimen versus those who received a Post-transplant Cyclophosphamide-based regimen?
* progression-free survival, Median overall survival, cumulative incidence of relapse, non-relapsed mortality (NRM) and GvHD at 2 years after Allo-SCT
* The impact of CMV infection and CMV reactivation on progression-free survival, overall survival, and NRM
* Averse events of GVHD prophylaxis medication Participants will be collected the data of treatment and treatment response during transplant until 2 years after transplant from hospital medical record.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 15 years
* Diagnosis of acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), chronic myeloid leukemia (CML), chronic lymphocytic leukemia (CLL), chronic myelomonocytic leukemia (CMML), myelodysplastic syndrome (MDS), myelofibrosis primary and/or post PV/ET myelofibrosis, aplastic anemia, lymphoma, or paroxysmal nocturnal hemoglobinuria
* Received HLA-matched related (MSD-HSCT) or unrelated allo-SCT (MUD-HSCT) or haploidentical hematopoietic stem cell transplantation

Exclusion Criteria:

* Insufficient data needed for analysis

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: allogeneic hematopoietic stem cell transplantation (allo-HSCT) patients
Sampling Method: Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with CMV infection and reactivation | 14 days to 6 months after transplant
  Number of participants with CMV infection and reactivation after allogeneic hematopoietic stem cell transplantation Between Standard Regimen, Methotrexate plus Cyclosporin A, and Post-transplant Cyclophosphamide-based Regimen

SECONDARY OUTCOMES:
progression-free survival | at 2 years after transplant
Median overall survival | at 2 years after transplant
cumulative incidence of relapse | at 2 years after transplant
non-relapsed mortality | at 2 years after transplant
GvHD | at 2 years after transplant
  Number of participants who have GvHD symptom
Averse events | at 2 years after transplant
  Averse events of GVHD prophylaxis medication

IPD SHARING:
Plan to Share IPD: Undecided
Need a consensus from colleagues